CLINICAL TRIAL: NCT06457711
Title: Blood Pressure and Cardiometabolic Risk in Postmenopausal Women With Hypertension and Obesity: A Real-World Study (Diet-to-HTN)
Brief Title: Blood Pressure and Cardiometabolic Risk (Diet-to-HTN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuliano Tocci, Associate Professor of Cardiology, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCTBPCMR
Record Dates: First submitted 2024-06-01; First posted 2024-06-13 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Arterial Hypertension; Menopause; Obesity; Cardiometabolic Syndrome; Cardiovascular Diseases
Keywords: blood pressure; diet; menopause; women; cardiometabolic risk
MeSH Terms: conditions — Hypertension; Obesity; Metabolic Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The investigators enrolled 50 patient to divide in 20 patients in the KD group, 20 in the IF group and 10 in the FD. Seven patients dropped out from their assigned groups as follows: FD (n = 2), IF (n = 3), and KD (n = 2).
Masking Description: Collaborative consultation encouraged patients to participate. Patient can choose their group of intervention. Dietary regimen were tailored on each patient: the intervention was adapted to patients' needs and to their body composition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Free diet Group (FDG) (Other): participants were offered nutritional guidance without strict limitations, but were encouraged to adhere to the principles of the Mediterranean diet and follow the dietary recommendations outlined in Harvard's Healthy Eating Plate.
  Interventions: Dietary Supplement: Free diet Group (FDG)
- Very low Calorie Ketogenic Diet Group (VLCKDG) (Experimental): the very low-calorie ketogenic diet (VLCKD) protocol involved limited carbohydrate consumption to less than 30 grams per day. The protocol suggested a protein intake ranging from 1 to 1.5 grams per kilogram of ideal body weight, with fats limited to 15-30 grams per day and total daily calories estimated between 600 and 800 kcal. During the initial three-week phase of the diet, participants replaced two meals per day with meal replacements-specifically, breakfast and one other main meal were substituted with a protein shake. Accompanying the shake for the main meal were low-glycemic-index vegetables in prescribed quantities.
  Interventions: Dietary Supplement: Very low Calorie Ketogenic Diet Group (VLCKDG)
- Intermittent Fasting Group (IFG) (Active Comparator): Our participant followed an intermittent fasting schedule, specifically the 16/8 method, which involves eating only during an eight-hour window each day and fasting for the subsequent sixteen hours. This eating period began at 12:00 noon and ended at 8:00 PM. During this window, the patient consumed three meals, each with a caloric value reduced by 25% from their total daily energy expenditure. The meals were based on the Mediterranean diet, focusing on the balance and quality of macronutrients.
  Interventions: Dietary Supplement: Intermittent Fasting Group (IFG)

INTERVENTIONS:
Dietary Supplement: Free diet Group (FDG) — Participants were offered nutritional guidance and were encouraged to adhere to the principles of the Mediterranean diet and follow the dietary recommendations outlined in Harvard's Healthy Eating Plate.
  Arms: Free diet Group (FDG)
Dietary Supplement: Very low Calorie Ketogenic Diet Group (VLCKDG) — Participants were offered nutritional guidance and were encouraged to adhere to the principles of the very low-calorie ketogenic diet (VLCKD) protocol
  Arms: Very low Calorie Ketogenic Diet Group (VLCKDG)
Dietary Supplement: Intermittent Fasting Group (IFG) — Participants were offered nutritional guidance and were encouraged to adhere to the principles of the intermittent fasting schedule
  Arms: Intermittent Fasting Group (IFG)

SUMMARY:
Obesity is a significant health issue that increases the risk of serious cardiovascular problems. In recent years, two dietary methods, the Ketogenic Diet (KD) and Intermittent Fasting (IF), have become popular for their potential to treat obesity and its related issue, hypertension. While both diets are known for their effectiveness in weight loss, their specific impacts on blood pressure (BP) and overall heart health risks are less understood especially in menopausal women.

The main goal of this study was to investigate how the Ketogenic Diet and Intermittent Fasting compare to a regular, unrestricted diet (referred to as Free Diet or FD) in terms of their effects on clinic blood pressure levels in menopausal women.

Additionally, the study looked at changes in Body Mass Index (BMI), the percentage of total body weight loss, body fat percentage, waist and hip measurements, the ratio of waist-to-hip size, and the Phase Angle (PhA), which is a measure of the body's overall health status.

DETAILED DESCRIPTION:
This research was conducted as a single-center, prospective, open-label clinical trial at Sant'Andrea Hospital in Rome, Italy. Participants included menopausal women with a BMI of 25 kg/m² or higher, who were already being treated for uncomplicated hypertension. These women were assessed at the hospital's Hypertension Unit and then placed into one of three diet groups: Ketogenic Diet, Intermittent Fasting, or Free Diet. Each participant received personalized dietary advice, underwent regular blood pressure checks aligned with European health guidelines, and completed standard health tests including electrocardiograms and blood tests for glucose, lipids, and liver and kidney functions. Measurements of all key health indicators were taken at the start of the study, then again after two months and six months.

This study is designed to offer clearer insights into how specific dietary choices can affect cardiovascular health and help manage hypertension in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* female individuals,
* aged between 50 and 65 years,
* BMI ≥25 kg/m2;
* diagnosis of essential uncomplicated arterial hypertension for at least 6 months;
* perimenopause or menopause confirmed,
* provision of informed consent.

Exclusion Criteria:

* previous history of major CVDs;
* severe heart or renal failure;
* poor adherence to prescribed pharmacological and non-pharmacological treatments;
* treated uncontrolled hypertension or diabetes;
* secondary forms of hypertension;
* uncontrolled thyroid diseases;
* previous bariatric surgery or endoscopic bariatric procedures;
* regular engagement in competitive sports activities;
* history of alcoholism and/or drug addiction;
* psychiatric and/or neurological conditions affecting the understanding and giving of informed consent;
* cancer or any other progressive severe disease;
* use of pharmacological treatments known to may interfere with the main purposes of the study protocol.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 50 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Clinic systolic brachial BP levels. | 6 months
  The primary aim was to evaluate the effects of Very low calorie Ketogenic Diet or intermittent fasting compared to Free Diet on clinic systolic brachial BP levels (mmHg).

SECONDARY OUTCOMES:
Body composition: BMI | 6 months
  Secondary outcomes included changes from baseline of Body Mass Index (BMI) weight and height will be combined to report BMI in kg/m^2.
Body composition: Fat mass (%) | 6 months
  Secondary outcomes included changes from baseline of Percentage of total body weight loss (TWL %), Body Fat Percentage (BFP %) derived from Bioelectrical impedance analysis (BIA)
Body composition: circumference | 6 months
  Secondary outcomes included changes from baseline of waist (WC) and hip circumference (cm), combined in waist-hip ratio (WHR)
Body Composition: Bioelectrical impedance analysis (BIA) | 6 months
  Secondary outcomes included changes from baseline of Phase Angle °
Clinic diastolic brachial BP levels. | 6 months
  Secondary outcomes included modulation of diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided